CLINICAL TRIAL: NCT02118792
Title: A Multicenter, Randomized, Double-Blind, Vehicle-Controlled Study of the Safety and Efficacy of AN2728 Topical Ointment, 2% in Children, Adolescents, and Adults (Ages 2 Years and Older) With Atopic Dermatitis
Brief Title: Safety and Efficacy of AN2728 Topical Ointment, 2% in Children, Adolescents, and Adults (Aged 2 Years and Older) With Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AN2728-AD-302
Record Dates: First submitted 2014-04-15; First posted 2014-04-21 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Dermatitis, Atopic
Keywords: atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AN2728 Topical Ointment, 2% (Experimental): AN2728 Topical Ointment, 2%, applied twice daily for up to 28 days
  Interventions: Drug: AN2728 Topical Ointment, 2%
- Matching vehicle control (Placebo Comparator): Matching vehicle control, applied twice daily for up to 28 days
  Interventions: Drug: Matching vehicle control

INTERVENTIONS:
Drug: AN2728 Topical Ointment, 2%
  Arms: AN2728 Topical Ointment, 2%
Drug: Matching vehicle control
  Arms: Matching vehicle control

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of AN2728 Topical Ointment, 2% in children, adolescents, and adults (ages 2 years and older) with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 2 years and older
* Has a clinical diagnosis of Atopic Dermatitis (AD) according to the criteria of Hanifin and Rajka
* Has AD involvement ≥ 5% Treatable %BSA (excluding the scalp)
* Has an ISGA score of Mild (2) or Moderate (3) at Baseline/Day 1
* All female subjects of childbearing potential must use acceptable methods of contraception from the Screening Visit continuously until 30 days after stopping study drug

Exclusion Criteria:

* As determined by the study doctor, a medical history that may interfere with study objectives
* Unstable AD or any consistent requirement for high potency topical corticosteroids
* History of use of biologic therapy (including intravenous immunoglobulin)
* Recent or anticipated concomitant use of systemic or topical therapies that might alter the course of AD
* Recent or current participation in another research study
* Females who are breastfeeding, pregnant, or with plans to get pregnant during the participation in the study
* Participation in a previous AN2728 clinical trial

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 764 (Actual)
Dates: Start 2014-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Anacor Investigational Site, Henrico, Virginia, United States

REFERENCES:
- [Derived] Stein Gold LF, Tom WL, Shi V, Sanders P, Zang C, Vlahos B, Cha A. Impact of Crisaborole in Treatment-Experienced Patients With Mild-to-Moderate Atopic Dermatitis. Dermatitis. 2024 Jan-Feb;35(1):84-91. doi: 10.1089/derm.2023.0112. Epub 2024 Jan 11. PMID 38206678
- [Derived] Luger TA, Hebert AA, Zaenglein AL, Silverberg JI, Tan H, Ports WC, Zielinski MA. Subgroup Analysis of Crisaborole for Mild-to-Moderate Atopic Dermatitis in Children Aged 2 to < 18 Years. Paediatr Drugs. 2022 Mar;24(2):175-183. doi: 10.1007/s40272-021-00490-y. Epub 2022 Mar 16. PMID 35292919
- [Derived] Geng B, Hebert AA, Takiya L, Miller L, Werth JL, Zang C, Sanders P, Lebwohl MG. Efficacy and Safety Trends with Continuous, Long-Term Crisaborole Use in Patients Aged >/= 2 Years with Mild-to-Moderate Atopic Dermatitis. Dermatol Ther (Heidelb). 2021 Oct;11(5):1667-1678. doi: 10.1007/s13555-021-00584-y. Epub 2021 Aug 11. PMID 34379285
- [Derived] Thyssen JP, Zang C, Neary MP, Bushmakin AG, Cappelleri JC, Cha A, Russo C, Luger TA. Translating the Investigator's Static Global Assessment to the Eczema Area and Severity Index in Studies of Crisaborole for Atopic Dermatitis. Dermatol Ther (Heidelb). 2021 Jun;11(3):845-853. doi: 10.1007/s13555-021-00509-9. Epub 2021 Mar 13. PMID 33728583
- [Derived] Stein Gold LF, Takiya L, Zang C, Sanders P, Feldman SR. Demographics and Baseline Disease Characteristics of Early Responders to Crisaborole for Atopic Dermatitis. J Drugs Dermatol. 2020 Jun 1;19(6):619-624. PMID 32574023
- [Derived] Silverberg JI, Tallman AM, Ports WC, Gerber RA, Tan H, Zielinski MA. Evaluating the Efficacy of Crisaborole Using the Atopic Dermatitis Severity Index and Percentage of Affected Body Surface Area. Acta Derm Venereol. 2020 Jun 11;100(13):adv00170. doi: 10.2340/00015555-3489. PMID 32318744
- [Derived] Simpson EL, Paller AS, Boguniewicz M, Eichenfield LF, Feldman SR, Silverberg JI, Chamlin SL, Zane LT. Crisaborole Ointment Improves Quality of Life of Patients with Mild to Moderate Atopic Dermatitis and Their Families. Dermatol Ther (Heidelb). 2018 Dec;8(4):605-619. doi: 10.1007/s13555-018-0263-0. Epub 2018 Oct 22. PMID 30345457
- [Derived] Paller AS, Tom WL, Lebwohl MG, Blumenthal RL, Boguniewicz M, Call RS, Eichenfield LF, Forsha DW, Rees WC, Simpson EL, Spellman MC, Stein Gold LF, Zaenglein AL, Hughes MH, Zane LT, Hebert AA. Efficacy and safety of crisaborole ointment, a novel, nonsteroidal phosphodiesterase 4 (PDE4) inhibitor for the topical treatment of atopic dermatitis (AD) in children and adults. J Am Acad Dermatol. 2016 Sep;75(3):494-503.e6. doi: 10.1016/j.jaad.2016.05.046. Epub 2016 Jul 11. PMID 27417017

RESULTS

PARTICIPANT FLOW:
Groups:
- AN2728 Ointment, 2 Percent (%): AN2728 ointment, 2% was applied topically twice daily, to all treatable atopic dermatitis (AD)-involved areas (excluding scalp), from Day 1 up to Day 28 in each participant. Treatable AD-involved areas were identified at Baseline (Day 1) by investigator.
- AN2728 Ointment, Vehicle: AN2728 ointment, vehicle was applied topically twice daily, to all treatable AD-involved areas (excluding scalp), from Day 1 up to Day 28 in each participant. Treatable AD-involved areas were identified at Baseline (Day 1) by investigator.
Period: Overall Study
Arm/Group | AN2728 Ointment, 2 Percent (%) | AN2728 Ointment, Vehicle
Started | 514 | 250
Treated | 513 | 250
Completed | 483 | 213
Not Completed | 31 | 37
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Lost to Follow-up | 4 | 4
Not completed — Adverse Event | 5 | 4
Not completed — Withdrawal by parent/guardian | 14 | 20
Not completed — Other | 1 | 6
Not completed — Randomised but not treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) population included all participants who were randomized and received study drug.
Groups:
- AN2728 Ointment, 2 Percent (%): AN2728 ointment, 2% was applied topically twice daily, to all treatable AD-involved areas (excluding scalp), from Day 1 up to Day 28 in each participant. Treatable AD-involved areas were identified at Baseline (Day 1) by investigator.
- Total: Total of all reporting groups
Arm/Group | AN2728 Ointment, 2 Percent (%) | AN2728 Ointment, Vehicle | Total
Number analyzed (Participants) | 513 | 250 | 763
Age, Customized [Count of Participants; unit: Participants]
  2 -11 years | 310 | 164 | 474
  12 -17 years | 126 | 57 | 183
  >=18 years | 77 | 29 | 106
Gender [Count of Participants; unit: Participants]
  Female | 282 | 138 | 420
  Male | 231 | 112 | 343

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Success in Investigator's Static Global Assessment (ISGA) Score at Day 29
Description: ISGA assessed the severity of AD (except scalp) on a 5-point scale ranged from 0 (clear) to 4 (maximum severe), where higher scores indicate higher degree of AD. Grades for classification of severity: 0= clear (minor residual hypo/hyper pigmentation, no erythema or induration or papulation, no oozing or crusting), 1= almost clear (trace faint pink erythema, with barely perceptible induration or papulation and no oozing or crusting), 2= mild (faint pink erythema with mild induration or papulation and no oozing or crusting), 3= moderate (pink-red erythema with moderate induration or papulation with or without oozing or crusting) and 4= severe (deep or bright red erythema with severe induration or papulation and with oozing or crusting). Treatment success was defined as an ISGA score of Clear (0) or Almost Clear (1) with at least a 2-grade improvement from baseline.
Time Frame: Day 29
Population: ITT population included all participants who were randomized and received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | AN2728 Ointment, 2 Percent (%) | AN2728 Ointment, Vehicle
Number analyzed (Participants) | 513 | 250
percentage of participants | 31.4 | 18.0
Statistical Analysis 1: Comparison: AN2728 Ointment, 2 Percent (%) vs AN2728 Ointment, Vehicle; Test type: Superiority or Other; p < 0.001, Regression, Logistic

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) And Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence attributed to a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; Initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug to the end of study, that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: AEs: Baseline (Day 1) up to Day 29, SAEs: Baseline (Day 1) up to Day 36
Population: Safety population included all randomized participants who had at least 1 confirmed dose of study drug, and had at least 1 post-baseline assessment.
Measure: Number; unit: participants
Arm/Group | AN2728 Ointment, 2 Percent (%) | AN2728 Ointment, Vehicle
Number analyzed (Participants) | 510 | 247
participants
  AEs | 150 | 79
  SAEs | 3 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Electrocardiogram (ECG) Findings at Day 8
Description: ECG parameters that were analyzed: PR interval, QRS interval, QT interval and corrected QT interval based on Fridericia's formula (QTcF). Clinical significance of change from baseline in ECG findings was determined by investigator.
Time Frame: Baseline, Day 8
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | AN2728 Ointment, 2 Percent (%) | AN2728 Ointment, Vehicle
Number analyzed (Participants) | 510 | 247
participants | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs at Day 36
Description: Following parameters were analyzed for examination of vital signs: systolic and diastolic blood pressure, pulse, respiratory rate and body temperature. Vital sign measurements were performed with the participant in the seated or supine position and after the participant had been calmly sitting or lying face up for a minimum of 5 minutes. Clinical significance of change from baseline value was determined by investigator.
Time Frame: Baseline (Day 1), Day 36
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | AN2728 Ointment, 2 Percent (%) | AN2728 Ointment, Vehicle
Number analyzed (Participants) | 510 | 247
participants | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Laboratory Values
Description: Laboratory values included: Alkaline Phosphatase, Alanine Aminotransferase, Aspartate Aminotransferase, Albumin, Bilirubin, Blood Urea Nitrogen, Glucose, Hematocrit, Hemoglobin, Leukocytes, Lymphocytes, Monocytes, Neutrophils, Platelets, Basophils, Eosinophils, Erythrocytes, Potassium, Protein, Sodium. Clinically significant laboratory abnormalities were defined as abnormal laboratory test values that have clinical manifestations or require medical intervention, as per investigator's discretion.
Time Frame: Baseline up to Day 36
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- AN2728 Topical Ointment, 2 Percent (%): AN2728 ointment, 2% was applied topically twice daily, to all treatable AD-involved areas (excluding scalp), from Day 1 up to Day 28 in each participant. Treatable AD-involved areas were identified at Baseline (Day 1) by investigator.
- AN2728 Topical Ointment, Vehicle: AN2728 ointment, vehicle was applied topically twice daily, to all treatable AD-involved areas (excluding scalp), from Day 1 up to Day 28 in each participant. Treatable AD-involved areas were identified at Baseline (Day 1) by investigator.
Arm/Group | AN2728 Topical Ointment, 2 Percent (%) | AN2728 Topical Ointment, Vehicle
Number analyzed (Participants) | 510 | 247
participants | 4 | 4

6. Primary Outcome: Percentage of Participants With Local Tolerability Symptoms at Baseline
Description: Local tolerability symptoms (burning/stinging) were assessed in participants at sites of study drug application. Symptoms were assessed on 4-point scale ranging from 0 to 3, where 0 = none (no stinging/burning), 1 = mild (slight warm, tingling sensation); 2= moderate (definite warm; tingling/stinging sensation that is somewhat bothersome and severe); 3= severe (hot, tingling/stinging sensation that caused definite discomfort). Higher scores indicated more severe symptoms. Percentage of participants with each level of local tolerability (none, mild, moderate, severe) symptoms were reported.
Time Frame: Baseline (Day 1)
Population: Safety population included all randomized participants who had at least 1 confirmed dose of study drug, and had at least 1 post-baseline assessment. Here, number of participants analyzed (N) signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | AN2728 Topical Ointment, 2 Percent (%) | AN2728 Topical Ointment, Vehicle
Number analyzed (Participants) | 509 | 247
percentage of participants
  None | 48.7 | 56.3
  Mild | 23.8 | 21.9
  Moderate | 19.6 | 16.6
  Severe | 7.9 | 5.3

7. Secondary Outcome: Percentage of Participants With an Investigator's Static Global Assessment (ISGA) Score of Clear (0) or Almost Clear (1) at Day 29
Description: ISGA assessed the severity of AD (except scalp and venous access area) on a 5-point scale ranged from 0 (clear) to 4 (maximum severe), where higher scores indicate higher degree of AD. Grades for classification of severity: 0= clear (minor residual discoloration, no erythema or induration or papulation, no oozing or crusting), 1= almost clear (trace faint pink erythema, with barely perceptible induration or papulation and no oozing or crusting), 2= mild (faint pink erythema with mild induration or papulation and no oozing or crusting), 3= moderate (pink-red erythema with moderate induration or papulation with or without oozing or crusting) and 4= severe (deep or bright red erythema with severe induration or papulation and with oozing or crusting). Percentage of participants with an ISGA score of 0 or 1 were reported.
Time Frame: Day 29
Population: ITT population included all participants who were randomized and received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | AN2728 Topical Ointment, 2 Percent (%) | AN2728 Topical Ointment, Vehicle
Number analyzed (Participants) | 513 | 250
percentage of participants | 48.5 | 29.7

8. Secondary Outcome: Time to Achieve Treatment Success Based on Investigator's Static Global Assessment (ISGA)
Description: Time to achieve treatment success based on ISGA was defined as the time interval between the administrations of first dose of study drug until first documentation of success in ISGA. Success in ISGA was defined as an ISGA score of clear (0) or almost clear (1) with at least 2-grade improvement from baseline. It was analyzed using Kaplan-Meier method.
Time Frame: Baseline up to Day 29
Population: ITT population included all participants who were randomized and received study drug.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | AN2728 Topical Ointment, 2 Percent (%) | AN2728 Topical Ointment, Vehicle
Number analyzed (Participants) | 513 | 250
days | NA [NA to NA] — The median time to achieve success in ISGA and its 95% confidence interval (CI) were not estimable, as fewer participants (less than 50 percent) reached success in ISGA. | NA [NA to NA] — The median time to achieve success in ISGA and its 95% CI were not estimable, as fewer participants (less than 50 percent) reached success in ISGA.

9. Secondary Outcome: Change From Baseline in Signs of Atopic Dermatitis at Day 29
Description: Signs of AD included erythema, induration/papulation, exudation, excoriation and lichenification. Each sign was assessed on a 4- point scale ranges from 0 to 3, where 0= none, 1= mild, 2= moderate to 3= severe. Higher score indicates severe signs and symptoms of AD.
Time Frame: Baseline, Day 29
Population: ITT population included all participants who were randomized and received study drug. Here, 'n' signifies those participants who were evaluable at specific time point for each arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AN2728 Topical Ointment, 2 Percent (%) | AN2728 Topical Ointment, Vehicle
Number analyzed (Participants) | 513 | 250
units on a scale
  Erythema: Baseline (n =513, 250) | 1.7 (0.59) | 1.6 (0.59)
  Erythema: Change at Day 29 (n =486, 224) | -0.7 (0.79) | -0.3 (0.81)
  Induration: Baseline (n =513, 250) | 1.8 (0.61) | 1.8 (0.56)
  Induration: Change at Day 29 (n =486, 224) | -0.7 (0.83) | -0.4 (0.76)
  Exudation: Baseline (n =513, 250) | 0.7 (0.78) | 0.6 (0.81)
  Exudation: Change at Day 29 (n =486, 224) | -0.4 (0.80) | -0.1 (0.84)
  Excoriation: Baseline (n =513, 250) | 1.5 (0.72) | 1.5 (0.68)
  Excoriation: Change at Day 29 (n =486, 224) | -0.7 (0.89) | -0.5 (0.93)
  Lichenification: Baseline (n =513, 250) | 1.5 (0.68) | 1.5 (0.76)
  Lichenification: Change at Day 29 (n =486, 224) | -0.6 (0.80) | -0.3 (0.76)

10. Other Pre Specified Outcome: Time to Improvement in Pruritus
Description: Time to improvement in pruritus was defined as the time interval between the administration of first dose of study drug till the first documentation of improvement in pruritus. Improvement in pruritus was defined as achieving none (0) or mild (1) score with at least a 1- grade improvement from baseline. Severity of pruritus was assessed on 4-point numeric scale ranges from 0 to 3, where 0= none (no itching), 1= mild (occasional, slight itching/scratching), 2= moderate (constant or intermittent itching/scratching which is not disturbing sleep) and 3= severe (bothersome itching/scratching which is disturbing sleep). Higher scores indicated more severe condition. It was analyzed using Kaplan-Meier method.
Time Frame: Baseline (Day 1) up to Day 29
Population: ITT population included all participants who were randomized and received study drug. Here, "N'' signifies those participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | AN2728 Topical Ointment, 2 Percent (%) | AN2728 Topical Ointment, Vehicle
Number analyzed (Participants) | 439 | 211
days | 1.41 [1.23 to 1.66] | 1.54 [1.20 to 1.93]

11. Other Pre Specified Outcome: Change From Baseline in Children's Dermatology Life Quality Index (CDLQI) Score at Day 29
Description: The CDLQI was a 10-item questionnaire that measures the impact of skin disease on children's (aged 2-15 years) quality of life. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicate more impact on quality of life. The CDLQI total score was the sum of individual scores of question 1-10 and ranges from 0 (not at all) to 30 (very much): 0-1 = no effect at all on the children's life; 2-6 = small effect on the children's life; 7-12 = moderate effect on the children's life; 13-18 = very large effect on the children's life; 19-30 = extremely large effect on the children's life. Higher scores indicate more impact on quality of life of children.
Time Frame: Baseline (Day 1), Day 29
Population: ITT population included all participants who were randomized and received study drug. Here, Number of participants analyzed (N) signifies those participants who were evaluable for this outcome measure and 'n' signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AN2728 Topical Ointment, 2 Percent (%) | AN2728 Topical Ointment, Vehicle
Number analyzed (Participants) | 404 | 204
units on a scale
  Baseline (n =404, 204) | 9.0 (5.77) | 8.9 (5.48)
  Change at Day 29 (n =376,180) | -4.0 (4.92) | -2.9 (5.01)

12. Other Pre Specified Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Score at Day 29
Description: The DLQI was a 10-item questionnaire that measures the impact of skin disease on participant's quality of life. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicate more impact on quality of life. The DLQI total score ranges from 0 (not at all) to 30 (very much): 0-1 = no effect at all on the participant's life; 2-6 = small effect on the participant's life; 7-12 = moderate effect on the participant's life; 13-18 = very large effect on the participant's life; 19-30 = extremely large effect on the participant's life. Higher scores indicate more impact on quality of life of participants.
Time Frame: Baseline (Day 1), Day 29
Population: ITT population included all participants who were randomized and received study drug. Here, ''N'' signifies those participants who were evaluable for this outcome measure and 'n' signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AN2728 Topical Ointment, 2 Percent (%) | AN2728 Topical Ointment, Vehicle
Number analyzed (Participants) | 97 | 40
units on a scale
  Baseline (n =97, 40) | 9.7 (6.24) | 9.1 (6.67)
  Change at Day 29 (n =93, 38) | -5.0 (5.49) | -3.4 (4.75)

13. Other Pre Specified Outcome: Change From Baseline in Dermatitis Family Impact Questionnaire (DFI) Score at Day 29
Description: The DFI was a 10-item disease questionnaire that measures the impact of having a child with AD on family quality of life. It was completed by parent/legal guardian of the child (affected by AD), based on recall over the past week. Each question was scored on a 4-point scale ranging from 0 (good) to 3 (worst), where higher scores indicated worst quality of life of family. The DFI total score was the sum of individual scores of the 10 questions and ranges from 0 (good) to 30 (worst), where higher DFI scores indicated worst quality of life of family.
Time Frame: Baseline (Day 1), Day 29
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AN2728 Topical Ointment, 2 Percent (%) | AN2728 Topical Ointment, Vehicle
Number analyzed (Participants) | 431 | 217
units on a scale
  Baseline (n =431, 217) | 7.7 (6.57) | 8.0 (5.65)
  Change at Day 29 (n =404, 190) | -3.6 (5.18) | -2.8 (4.75)

14. Primary Outcome: Percentage of Participants With Local Tolerability Symptoms at Day 8
Description: Local tolerability symptoms (burning/stinging) were assessed in participants at sites of study drug application. Symptoms were assessed on 4-point scale ranging from 0 to 3, where 0= none (no stinging/burning), 1 = mild (slight warm, tingling sensation); 2= moderate (definite warm; tingling/stinging sensation that is somewhat bothersome and severe); 3= severe (hot, tingling/stinging sensation that caused definite discomfort). Higher scores indicated more severe symptoms. Percentage of participants with each level of local tolerability (none, mild, moderate, severe) symptoms were reported.
Time Frame: Day 8
Population: Safety population included all randomized participants who had at least 1 confirmed dose of study drug, and had at least 1 post-baseline assessment. Here, "N" signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | AN2728 Topical Ointment, 2 Percent (%) | AN2728 Topical Ointment, Vehicle
Number analyzed (Participants) | 508 | 244
percentage of participants
  None | 63.8 | 73.0
  Mild | 24.0 | 14.8
  Moderate | 9.1 | 11.5
  Severe | 3.1 | 0.8

15. Primary Outcome: Percentage of Participants With Local Tolerability Symptoms at Day 15
Description: Local tolerability symptoms (burning/stinging) were assessed in participants at sites of study drug application. Symptoms were assessed on 4-point scale ranging from 0 to 3, where 0= none (no stinging/burning), 1= mild (slight warm, tingling sensation); 2= moderate (definite warm; tingling/stinging sensation that is somewhat bothersome and severe); 3= severe (hot, tingling/stinging sensation that caused definite discomfort). Higher scores indicated more severe symptoms. Percentage of participants with each level of local tolerability (none, mild, moderate, severe) symptoms were reported.
Time Frame: Day 15
Population: Safety population included all randomized participants who had at least 1 confirmed dose of study drug, and had at least 1 post-baseline assessment. Here, "N" signifies those participants who were analyzed in this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | AN2728 Topical Ointment, 2 Percent (%) | AN2728 Topical Ointment, Vehicle
Number analyzed (Participants) | 488 | 239
percentage of participants
  None | 68.0 | 70.7
  Mild | 20.9 | 15.5
  Moderate | 7.4 | 9.6
  Severe | 3.7 | 4.2

16. Primary Outcome: Percentage of Participants With Local Tolerability Symptoms at Day 22
Description: Local tolerability symptoms (burning/stinging) were assessed in participants at sites of study drug application. Symptoms were assessed on 4-point scale which ranges from 0 to 3, where 0 = none (no stinging/burning), 1 = mild (slight warm, tingling sensation); 2= moderate (definite warm; tingling/stinging sensation that is somewhat bothersome and severe); 3= severe (hot, tingling/stinging sensation that caused definite discomfort). Higher scores indicate high severity of symptoms. In this outcome, percentage of participants with each level of local tolerability (none, mild, moderate, severe) symptoms were reported.
Time Frame: Day 22
Population: Safety population included all randomized participants who had at least 1 confirmed dose of study drug, and had at least 1 post-baseline assessment. Here, number of participants analyzed "N" signifies those participants who were analyzed in this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | AN2728 Topical Ointment, 2 Percent (%) | AN2728 Topical Ointment, Vehicle
Number analyzed (Participants) | 487 | 227
percentage of participants
  None | 69.0 | 71.4
  Mild | 21.8 | 16.7
  Moderate | 6.8 | 8.4
  Severe | 2.5 | 3.5

17. Primary Outcome: Percentage of Participants With Local Tolerability Symptoms at Day 29
Description: Local tolerability symptoms (burning/stinging) were assessed in participants at sites of study drug application. Symptoms were assessed on 4-point scale which ranges from 0 to 3, where 0 = none (no stinging/burning), 1 = mild (slight warm, tingling sensation); 2= moderate (definite warm; tingling/stinging sensation that is somewhat bothersome and severe); 3= severe (hot, tingling/stinging sensation that caused definite discomfort). Higher scores indicate high severity of symptoms. Percentage of participants with each level of local tolerability (none, mild, moderate, severe) symptoms were reported.
Time Frame: Day 29
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | AN2728 Topical Ointment, 2 Percent (%) | AN2728 Topical Ointment, Vehicle
Number analyzed (Participants) | 486 | 222
percentage of participants
  None | 70.4 | 73.9
  Mild | 17.3 | 13.5
  Moderate | 10.1 | 10.8
  Severe | 2.3 | 1.8

18. Primary Outcome: Percentage of Participants With Local Tolerability Symptoms at Day 36
Description: as for outcome 17
Time Frame: Day 36
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | AN2728 Topical Ointment, 2 Percent (%) | AN2728 Topical Ointment, Vehicle
Number analyzed (Participants) | 474 | 213
percentage of participants
  None | 71.1 | 77.5
  Mild | 14.3 | 9.9
  Moderate | 9.1 | 10.3
  Severe | 5.5 | 2.3

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. AEs and SAEs were analyzed for safety population which included all randomized participants who received at least 1 confirmed dose of study drug, and had at least 1 post-baseline assessment.
Groups:
- AN2728 Topical Ointment, 2 Percent (%): AN2728 ointment 2% was applied topically twice daily, to all treatable AD-involved areas (excluding scalp), from Day 1 up to Day 28 in each participant. Treatable AD-involved areas were identified at Baseline (Day 1) by investigator.
- AN2728 Topical Ointment, Vehicle: AN2728 ointment vehicle was applied topically twice daily, to all treatable AD-involved areas (excluding scalp), from Day 1 up to Day 28 in each participant. Treatable AD-involved areas were identified at Baseline (Day 1) by investigator.
Arm/Group | AN2728 Topical Ointment, 2 Percent (%) | AN2728 Topical Ointment, Vehicle
Serious Adverse Events (participants affected / at risk) | 3/510 | 0/247
Other Adverse Events (participants affected / at risk) | 92/510 | 54/247
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AN2728 Topical Ointment, 2 Percent (%) (N=510) | AN2728 Topical Ointment, Vehicle (N=247)
Application site infection (Infections and infestations) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AN2728 Topical Ointment, 2 Percent (%) (N=510) | AN2728 Topical Ointment, Vehicle (N=247)
Diarrhoea (Gastrointestinal disorders) | 6 | 2
Vomiting (Gastrointestinal disorders) | 7 | 2
Application site pain (General disorders) | 14 | 3
Application site pruritus (General disorders) | 1 | 3
Application site urticaria (General disorders) | 0 | 3
Pyrexia (General disorders) | 7 | 4
Nasopharyngitis (Infections and infestations) | 9 | 6
Staphylococcal skin infection (Infections and infestations) | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 16 | 5
Headache (Nervous system disorders) | 6 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 4 | 6
Eczema (Skin and subcutaneous tissue disorders) | 3 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.